CLINICAL TRIAL: NCT00394914
Title: A Placebo-Controlled Study of the Effects of Pleconaril Nasal Spray on Common Cold Symptoms and Asthma Exacerbations Following Rhinovirus Exposure
Brief Title: Effects of Pleconaril Nasal Spray on Common Cold Symptoms and Asthma Exacerbations Following Rhinovirus Exposure (Study P04295)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: P04295; Doc ID: 3303796
Record Dates: First submitted 2006-10-31; First posted 2006-11-02 (Estimated); Results first posted 2013-10-31 (Estimated); Last update posted 2015-07-16 (Estimated); Status verified 2015-06

CONDITIONS: Asthma; Common Cold; Picornavirus Infection; Rhinovirus
MeSH Terms: conditions — Asthma; Common Cold; Picornaviridae Infections | interventions — pleconaril

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pleconaril (Experimental): Participants will receive Pleconaril nasal spray 4 sprays per nostril twice daily (BID), 24 mg/day for 1 week during the Treatment Period for a total of 14 doses.
  Interventions: Drug: Pleconaril
- Placebo (Placebo Comparator): Participants will receive placebo nasal spray 4 sprays per nostril BID for 1 week during the Treatment Period for a total of 14 doses.
  Interventions: Drug: Placebo to Pleconaril

INTERVENTIONS:
Drug: Pleconaril — Pleconaril nasal suspension is supplied in a bottle containing 120 actuations. Each actuation contains 1.5 mg of pleconaril.
  Other Names: SCH 900819
  Arms: Pleconaril
Drug: Placebo to Pleconaril — Placebo nasal suspension
  Arms: Placebo

SUMMARY:
This is a randomized, multi-center, double-blind, placebo-controlled study evaluating the efficacy of pleconaril nasal spray in preventing asthma exacerbation and common cold symptoms in asthmatic participants exposed to picornavirus respiratory infections. Participants will be assigned treatment with pleconaril or placebo nasal spray for 7 days (14 doses). Participants will be followed for an additional 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Must be ≥6 to ≤65 years of age, of either sex, and of any race, with a diagnosis of asthma at least 2 years prior to the Screening Visit.
* Must have a history of two or more upper respiratory infection-induced asthma exacerbations in the past 24 months.

  * For participants 6 to 17 years of age, exacerbations for the purpose of the inclusion criteria, will be defined as:
  * An increase of four or more puffs of a short-acting beta-agonist (SABA) per day for at least 3 consecutive days, or
  * An increase of two or more nebulizations of a SABA per day for at least 3 consecutive days, or
  * Documentation of morning (AM) peak flow drops >20% per day for at least 2 consecutive days, or
  * Documentation of AM peak flow drops of ≥50% for at least 1 day.
* Must have been on a stable dose of any asthma medication (including immunotherapy) for at least 1 month prior to the Screening Visit.
* Must have a pre-bronchodilator FEV1 ≥50% predicted at the Screening Visit, when all prohibited medications have been withheld for the specified interval.
* If a reversibility test has not been performed within the previous 24 months, a participant, ≥17 years of age, must demonstrate an increase in absolute FEV1 of ≥12%, with an absolute volume increase of at least 200 mL. A participant <17 years of age, must demonstrate an increase in absolute FEV1 ≥12%.
* Must cohabit with at least one other person (family member, roommate).
* A participant (or the participant's legal representation) must be willing to give written informed consent and be able to adhere to dose and visit schedules.
* Must be free of any clinically significant disease, other than asthma, which would interfere with study evaluation.
* Must be in general good health, as confirmed by routine clinical and laboratory testing. All laboratory tests (Complete Blood Count, blood chemistries, and urinalysis) and elctrocardiograms must be within normal limits or clinically acceptable to the investigator/sponsor.
* Female of childbearing potential must be using a medically acceptable, adequate form of birth control.

Exclusion Criteria:

* Had an upper or lower respiratory illness or exhibits signs and/or symptoms of a respiratory illness in the 4 weeks prior to the Screening Visit.
* Received any treatment more recently than the indicated washout period prior to Screening or who must continue to receive treatment that is prohibited.
* Smoker or ex-smoker and has smoked within the previous 5 years of Screening or has had a cumulative smoking history >10 pack years.
* Allergy/sensitivity to the study drug or its excipients.
* Female who is breast-feeding, pregnant, or intends to become pregnant.
* Used any investigational drugs within 30 days of Screening.
* Participating in any other clinical study.
* Part of the staff personnel directly involved with this study.
* Family member of the investigational study staff.

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 311 (Actual)
Dates: Start 2006-08; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All enrolled participants were screened. After the screening visit and before randomization, participants received weekly phone calls and revisited the site once per month during a Pre-exposure Period until exposed to a household member with a cold (index case).
Groups:
- All Participants (Pre-randomization): All participants on study prior to randomization.
- Pleconaril: Participants were randomized to receive Pleconaril nasal spray 4 sprays per nostril twice daily (BID), 24 mg/day for 1 week during the Treatment Period for a total of 14 doses.
- Placebo: Participants were randomized to receive placebo nasal spray 4 sprays per nostril BID for 1 week during the Treatment Period for a total of 14 doses.
Period: Screening Period
Arm/Group | All Participants (Pre-randomization) | Pleconaril | Placebo
Started | 311 | 0 | 0
Completed | 311 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Pre-exposure Period
Arm/Group | All Participants (Pre-randomization) | Pleconaril | Placebo
Started | 311 | 0 | 0
Completed | 311 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Treatment Period
Arm/Group | All Participants (Pre-randomization) | Pleconaril | Placebo
Started | 0 | 154 | 157
Completed | 0 | 144 | 151
Not Completed | 0 | 10 | 6
Not completed — Adverse Event | 0 | 3 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 2
Not completed — Noncompliance with protocol | 0 | 3 | 2
Not completed — Did not meet protocol eligibility | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Pleconaril: Participants received Pleconaril nasal spray 4 sprays per nostril twice daily (BID), 24 mg/day for 1 week during the Treatment Period for a total of 14 doses.
- Placebo: Participants received placebo nasal spray 4 sprays per nostril BID for 1 week during the Treatment Period for a total of 14 doses.
- Total: Total of all reporting groups
Arm/Group | Pleconaril | Placebo | Total
Number analyzed (Participants) | 154 | 157 | 311
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.4 (16.7) | 28.7 (17.3) | 29.1 (17.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85 | 97 | 182
  Male | 69 | 60 | 129

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Rhinovirus PCR-Positive Colds
Description: The common cold was defined as moderate or severe rhinorrhea and at least one other cold symptom of moderate to severe intensity for at least 1 day, together with rhinovirus-positive polymerase chain reaction (PCR), after a participant had temporal exposure to an index case. PCR+ was defined as positive or equivocal outcome of the picornavirus test any time after randomization.
Time Frame: From time of exposure to index case to end of Follow-up Period (21 days)
Population: Efficacy analyses were based on all randomized participants (intent-to-treat principle) with at least some follow-up information. Randomized participants with no follow-up information were included in the number of participants assigned to each treatment group to determine rhinovirus cold.
Measure: Number; unit: percentage of participants
Arm/Group | Pleconaril | Placebo
Number analyzed (Participants) | 154 | 157
percentage of participants | 2.6 | 2.5
Statistical Analysis 1: Comparison: Pleconaril vs Placebo; Test type: Superiority or Other; p = 0.973, Cochran-Mantel-Haenszel

2. Primary Outcome: Percentage of Participants With Asthma Exacerbations Together With Rhinovirus-Positive PCR
Description: Asthma exacerbation was defined as a participant having one of the following:
  1. 0.5 point or more increase in the Asthma Control Questionnaire (ACQ) from Baseline at Day 7. The ACQ is a validated instrument containing 7 questions to assess asthma control which incorporates symptoms, beta-agonist use, and spirometry. Participants recall their experiences during the previous 7 days and respond to each question using a 7-point scale. The items are equally weighted and the ACQ score is the mean of the 7 items and therefore ranges between 0 (well controlled) and 6 (extremely poorly controlled). The ACQ completed on the day of exposure was the Baseline ACQ.
  2. Any change to asthma treatment as prescribed by a physician, unscheduled contact (either office visit or phone contact where medication was changed for asthma symptoms), emergency room visit, or hospitalization.
  PCR+ was defined as positive or equivocal outcome of the picornavirus test any time after randomization.
Time Frame: From time of exposure to index case to end of Follow-up Period (21 days)
Population: Efficacy analyses were based on all randomized participants (intent-to-treat principle) with at least some follow-up information. Randomized participants with no follow-up information were included in the number of participants assigned to each treatment group to determine exacerbation.
Measure: Number; unit: percentage of participants
Arm/Group | Pleconaril | Placebo
Number analyzed (Participants) | 154 | 157
percentage of participants | 1.3 | 2.5
Statistical Analysis 1: Comparison: Pleconaril vs Placebo; Test type: Superiority or Other; p = 0.425, Cochran-Mantel-Haenszel

3. Secondary Outcome: LS Mean Change From Baseline in the Asthma Control Questionnaire (ACQ)
Description: The ACQ is a validated instrument containing 7 questions to assess asthma control which incorporates symptoms, beta-agonist use, and spirometry. Participants recall their experiences during the previous 7 days and respond to each question using a 7-point scale. The items are equally weighted and the ACQ score is the mean of the 7 items and therefore ranges between 0 (well controlled) and 6 (extremely poorly controlled). The ACQ completed on the day of exposure was the Baseline ACQ. Pooled standard deviations (SDs) and least square (LS) means were calculated based on an analysis of variates (ANOVA) model.
Time Frame: Baseline through the Final Visit (Day 21)
Population: Efficacy analyses were based on all randomized participants (intent-to-treat principle) with at least some ACQ follow-up information.
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pleconaril | Placebo
Number analyzed (Participants) | 126 | 127
units on a scale
  Baseline (n=126, n=127) | 0.86 (0.72) | 0.87 (0.72)
  Change From BL to Day 8 (n=120, n=124) | -0.11 (0.52) | -0.06 (0.52)
  Change From BL to Day 14 (n=94, n=96) | -0.09 (0.58) | -0.15 (0.58)
  Change From BL to Day 21 (n=89, n=96) | -0.12 (0.56) | -0.02 (0.56)
  Change From BL to Final Visit (n=126, n=127) | -0.09 (0.56) | -0.00 (0.56)

4. Secondary Outcome: LS Mean Change From Baseline in Forced Expiratory Volume in 1 Second (FEV1)
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration. Pooled SDs and LS means were calculated based on an ANOVA model.
Time Frame: Baseline through the Final Visit (Day 21)
Population: Efficacy analyses were based on all randomized participants (intent-to-treat principle) with at least some FEV1 follow-up information.
Measure: Least Squares Mean (Standard Deviation); unit: liters
Arm/Group | Pleconaril | Placebo
Number analyzed (Participants) | 152 | 156
liters
  Baseline (n=152, n=156) | 2.335 (0.728) | 2.214 (0.728)
  Change From BL to Day 2 (n=111, n=115) | -0.091 (0.267) | -0.100 (0.267)
  Change From BL to Day 4 (n=97, n=102) | -0.059 (0.273) | -0.141 (0.273)
  Change From BL to Day 8 (n=132, n=135) | -0.070 (0.274) | -0.121 (0.274)
  Change From BL to Day 10 (n=116, n=120) | -0.090 (0.271) | -0.109 (0.271)
  Change From BL to Day 14 (n=140, n=139) | -0.063 (0.266) | -0.090 (0.266)
  Change From BL to Day 21 (n=141, n=146) | -0.080 (0.287) | -0.133 (0.287)
  Change From BL to Final Visit (n=152, n=156) | -0.076 (0.291) | -0.141 (0.291)

5. Secondary Outcome: LS Mean Change From Baseline in Peak Expiratory Flow (PEF) in AM
Description: PEF is a person's maximum speed of expiration as measured with a peak flow meter and was measured twice daily in the morning (AM) and evening (PM). Pooled SDs and LS means were calculated based on an ANOVA model.
Time Frame: Baseline through the Final Visit (Day 21)
Population: Efficacy analyses were based on all randomized participants (intent-to-treat principle) with at least some PEF follow-up information.
Measure: Least Squares Mean (Standard Deviation); unit: L/min
Arm/Group | Pleconaril | Placebo
Number analyzed (Participants) | 124 | 136
L/min
  Baseline (n=124, n=136) | 306.2 (96.8) | 284.0 (96.8)
  Change From BL to Day 2 (n=108, n=123) | -0.1 (55.4) | -1.9 (55.4)
  Change From BL to Day 3 (n=103, n=120) | 9.9 (57.7) | 6.1 (57.7)
  Change From BL to Day 4 (n=103, n=118) | 5.1 (59.1) | -1.1 (59.1)
  Change From BL to Day 5 (n=96, n=122) | 0.2 (45.9) | -3.4 (45.9)
  Change From BL to Day 6 (n=104, n=114) | 0.2 (60.3) | 2.5 (60.3)
  Change From BL to Day 7 (n=102, n=112) | 2.5 (57.5) | -4.0 (57.5)
  Change From BL to Day 8 (n=102, n=116) | -0.6 (47.0) | -0.9 (47.0)
  Change From BL to Day 9 (n=105, n=114) | 13.6 (63.9) | 8.1 (63.9)
  Change From BL to Day 10 (n=90, n=102) | 7.7 (54.6) | 0.6 (54.6)
  Change From BL to Day 11 (n=95, n=108) | -3.9 (51.4) | -0.6 (51.4)
  Change From BL to Day 12 (n=94, n=102) | 3.2 (77.8) | 11.5 (77.8)
  Change From BL to Day 13 (n=88, n=97) | 4.7 (55.3) | 7.7 (55.3)
  Change From BL to Day 14 (n=90, n=103) | 3.4 (69.3) | 23.5 (69.3)
  Change From BL to Day 15 (n=91, n=107) | -3.2 (76.8) | 3.9 (76.8)
  Change From BL to Day 16 (n=92, n=101) | 4.4 (49.5) | -1.7 (49.5)
  Change From BL to Day 17 (n=74, n=93) | 6.0 (51.0) | -6.9 (51.0)
  Change From BL to Day 18 (n=80, n=98) | 0.7 (57.9) | 10.8 (57.9)
  Change From BL to Day 19 (n=81, n=102) | 1.2 (62.7) | 4.1 (62.7)
  Change From BL to Day 20 (n=76, n=88) | 10.2 (58.0) | 10.4 (58.0)
  Change From BL to Day 21 (n=62, n=85) | 10.5 (49.1) | -1.4 (49.1)
  Change From BL to Final Day (n=124, n=136) | 4.6 (57.8) | -5.2 (57.8)
  Change From BL to Week 1 (n=122, n=136) | -0.7 (39.2) | -2.2 (39.2)
  Change From BL to Week 2 (n=119, n=134) | 1.4 (45.9) | 4.5 (45.9)
  Change From BL to Week 3 (n=109, n=127) | 5.2 (48.7) | -1.1 (48.7)
  Change From BL to Final Week (n=124, n=136) | 2.3 (49.8) | -3.8 (49.8)

6. Secondary Outcome: LS Mean Change From Baseline in Peak Expiratory Flow (PEF) in PM
Description: as for outcome 5
Time Frame: Baseline through the Final Visit (Day 21)
Population: as for outcome 5
Measure: Least Squares Mean (Standard Deviation); unit: L/min
Arm/Group | Pleconaril | Placebo
Number analyzed (Participants) | 119 | 128
L/min
  Baseline (n=119, n=128) | 310.9 (93.6) | 293.4 (93.6)
  Change From BL to Day 1 (n=93, n=105) | 0.4 (48.2) | 1.0 (48.2)
  Change From BL to Day 2 (n=102, n=115) | 2.0 (57.7) | 0.4 (57.7)
  Change From BL to Day 3 (n=98, n=112) | 2.3 (45.6) | -14.7 (45.6)
  Change From BL to Day 4 (n=98, n=108) | 8.2 (54.2) | 3.1 (54.2)
  Change From BL to Day 5 (n=105, n=109) | -3.7 (57.0) | 1.6 (57.0)
  Change From BL to Day 6 (n=98, n=108) | -3.5 (46.3) | -9.8 (46.3)
  Change From BL to Day 7 (n=95, n=106) | 10.0 (59.1) | -1.6 (59.1)
  Change From BL to Day 8 (n=94, n=106) | 11.2 (76.7) | 20.2 (76.7)
  Change From BL to Day 9 (n=91, n=103) | 3.5 (52.6) | -3.4 (52.6)
  Change From BL to Day 10 (n=91, n=99) | 9.2 (58.9) | 9.1 (58.9)
  Change From BL to Day 11 (n=83, n=97) | -3.0 (62.7) | 1.0 (62.7)
  Change From BL to Day 12 (n=82, n=90) | -2.6 (71.5) | 8.9 (71.5)
  Change From BL to Day 13 (n=85, n=98) | 9.3 (56.4) | 8.1 (56.4)
  Change From BL to Day 14 (n=80, n=98) | 2.4 (48.6) | 1.7 (48.6)
  Change From BL to Day 15 (n=88, n=89) | -0.2 (49.7) | -9.0 (49.7)
  Change From BL to Day 16 (n=82, n=84) | -6.8 (49.4) | -6.1 (49.4)
  Change From BL to Day 17 (n=81, n=93) | -1.1 (54.8) | -1.1 (54.8)
  Change From BL to Day 18 (n=84, n=97) | 3.2 (59.4) | 3.7 (59.4)
  Change From BL to Day 19 (n=80, n=93) | -1.0 (55.8) | 12.3 (55.8)
  Change From BL to Day 20 (n=78, n=80) | 16.2 (64.8) | 12.6 (64.8)
  Change From BL to Day 21 (n=47, n=63) | -7.5 (96.1) | 12.3 (96.1)
  Change From BL to Final Day (n=119, n=128) | 10.4 (81.1) | 14.7 (81.1)
  Change From BL to Week 1 (n=116, n=127) | 2.5 (38.4) | -2.0 (38.4)
  Change From BL to Week 2 (n=113, n=124) | 3.4 (49.2) | 6.0 (49.2)
  Change From BL to Week 3 (n=103, n=117) | -3.5 (49.5) | 3.5 (49.5)
  Change From BL to Final Week (n=119, n=128) | 3.1 (53.6) | 8.1 (53.6)

7. Secondary Outcome: LS Mean Change From Baseline in Total Cold Symptom Score
Description: Participants entered their cold symptoms into an e-diary twice daily beginning at the Screening Visit through completion of the study. The total cold symptom score was the sum of 6 scores for rhinorrhea, nasal congestion, cough, score throat, malaise, and myalgia. Each symptom is scored as follows: 0 = none-sign/symptom is not present, 1 = mild-sign/symptom noticeable but did not bother me or interfere with my normal daily activities/sleep, 2 = moderate- sign/symptom annoying and may have interfered with my normal daily activities/sleep, or 3 = severe-symptom very uncomfortable and interfered with most or all of my normal daily activities/sleep. The total score ranges from 0 to 18, with increasing scores reflecting more severe colds. Baseline values were defined as the average of the last seven assessments prior to randomization (before exposure to an index case). Pooled SDs and LS means were calculated based on an ANOVA model.
Time Frame: Baseline through the Final Visit (Day 21)
Population: Efficacy analyses were based on all randomized participants (intent-to-treat principle) with at least some cold symptom score follow-up information.
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pleconaril | Placebo
Number analyzed (Participants) | 147 | 153
units on a scale
  Baseline (n=147, n=153) | 1.09 (1.62) | 0.99 (1.62)
  Change From BL to Day 1 (n=135, n=143) | 0.03 (1.05) | 0.12 (1.05)
  Change From BL to Day 2 (n=143, n=152) | 0.21 (1.08) | 0.26 (1.08)
  Change From BL to Day 3 (n=141, n=152) | 0.31 (1.34) | 0.35 (1.34)
  Change From BL to Day 4 (n=142, n=152) | 0.14 (1.41) | 0.39 (1.41)
  Change From BL to Day 5 (n=140, n=152) | 0.04 (1.43) | 0.45 (1.43)
  Change From BL to Day 6 (n=136, n=152) | -0.01 (1.51) | 0.40 (1.51)
  Change From BL to Day 7 (n=139, n=150) | 0.03 (1.65) | 0.38 (1.65)
  Change From BL to Day 8 (n=139, n=149) | 0.02 (1.63) | 0.34 (1.63)
  Change From BL to Day 9 (n=138, n=150) | 0.04 (1.63) | 0.29 (1.63)
  Change From BL to Day 10 (n=139, n=150) | 0.18 (1.71) | 0.29 (1.71)
  Change From BL to Day 11 (n=137, n=149) | 0.17 (1.81) | 0.31 (1.81)
  Change From BL to Day 12 (n=137, n=148) | 0.07 (1.77) | 0.25 (1.77)
  Change From BL to Day 13 (n=136, n=146) | -0.02 (1.66) | 0.11 (1.66)
  Change From BL to Day 14 (n=138, n=146) | 0.05 (1.51) | 0.15 (1.51)
  Change From BL to Day 15 (n=135, n=144) | 0.04 (1.65) | 0.18 (1.65)
  Change From BL to Day 16 (n=132, n=144) | 0.04 (1.71) | 0.21 (1.71)
  Change From BL to Day 17 (n=133, n=145) | -0.06 (1.52) | 0.10 (1.52)
  Change From BL to Day 18 (n=137, n=146) | -0.17 (1.64) | -0.03 (1.64)
  Change From BL to Day 19 (n=132, n=145) | -0.03 (1.74) | -0.04 (1.74)
  Change From BL to Day 20 (n=126, n=136) | -0.04 (1.63) | 0.17 (1.63)
  Change From BL to Day 21 (n=108, n=121) | 0.15 (1.44) | 0.29 (1.44)
  Change From BL to Final Day (n=147, n=153) | 0.18 (1.58) | 0.23 (1.58)

8. Secondary Outcome: LS Mean Change From Baseline in Total Asthma Symptom Score
Description: Participants entered their asthma symptoms into an e-diary twice daily beginning at the Screening Visit through completion of the study. The total asthma symptom score was the sum of 3 scores for wheeze, cough, and dyspnea. Each symptom is scored as follows: 0 = none-sign/symptom is not present, 1 = mild-sign/symptom noticeable but did not bother me or interfere with my normal daily activities/sleep, 2 = moderate- sign/symptom annoying and may have interfered with my normal daily activities/sleep, or 3 = severe-symptom very uncomfortable and interfered with most or all of my normal daily activities/sleep. The total score ranges from 0 to 9, with increasing scores reflecting more severe asthma. Baseline values were defined as the average of the last seven assessments prior to randomization (before exposure to an index case). Pooled SDs and LS means were calculated based on an ANOVA model.
Time Frame: Baseline through the Final Visit (Day 21)
Population: Efficacy analyses were based on all randomized participants (intent-to-treat principle) with at least some asthma symptom score follow-up information.
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pleconaril | Placebo
Number analyzed (Participants) | 147 | 153
units on a scale
  Baseline (n=147, n=153) | 0.67 (1.03) | 0.56 (1.03)
  Change From BL to Day 1 (n=135, n=143) | 0.02 (0.71) | 0.08 (0.71)
  Change From BL to Day 2 (n=143, n=152) | 0.05 (0.60) | 0.07 (0.60)
  Change From BL to Day 3 (n=141, n=152) | 0.04 (0.65) | 0.09 (0.65)
  Change From BL to Day 4 (n=142, n=152) | -0.04 (0.77) | 0.09 (0.77)
  Change From BL to Day 5 (n=140, n=152) | -0.10 (0.81) | 0.15 (0.81)
  Change From BL to Day 6 (n=136, n=152) | -0.10 (0.88) | 0.15 (0.88)
  Change From BL to Day 7 (n=139, n=150) | -0.07 (0.90) | 0.18 (0.90)
  Change From BL to Day 8 (n=139, n=149) | -0.07 (0.95) | 0.12 (0.95)
  Change From BL to Day 9 (n=138, n=150) | -0.07 (0.88) | 0.10 (0.88)
  Change From BL to Day 10 (n=139, n=150) | -0.01 (0.96) | 0.15 (0.96)
  Change From BL to Day 11 (n=137, n=149) | -0.05 (1.02) | 0.17 (1.02)
  Change From BL to Day 12 (n=137, n=148) | -0.02 (1.02) | 0.09 (1.02)
  Change From BL to Day 13 (n=136, n=146) | -0.06 (0.92) | 0.02 (0.92)
  Change From BL to Day 14 (n=138, n=146) | -0.07 (0.85) | 0.03 (0.85)
  Change From BL to Day 15 (n=135, n=144) | -0.11 (0.86) | 0.08 (0.86)
  Change From BL to Day 16 (n=132, n=144) | -0.16 (0.93) | 0.04 (0.93)
  Change From BL to Day 17 (n=133, n=145) | -0.18 (0.84) | 0.00 (0.84)
  Change From BL to Day 18 (n=137, n=146) | -0.14 (0.91) | -0.05 (0.91)
  Change From BL to Day 19 (n=132, n=145) | -0.14 (1.03) | -0.04 (1.03)
  Change From BL to Day 20 (n=126, n=136) | -0.15 (0.97) | -0.01 (0.97)
  Change From BL to Day 21 (n=108, n=121) | -0.10 (0.93) | 0.06 (0.93)
  Change From BL to Final Day (n=147, n=153) | -0.09 (0.94) | 0.03 (0.94)

9. Secondary Outcome: LS Mean Change From Baseline in Short-acting Beta-Agonist (SABA) Rescue Medication Usage
Description: SABAs such as albuterol were permitted during the study as rescue medication and required a 6-hour washout prior to each visit. Participants entered their asthma medication use into an e-diary twice daily beginning at the Screening Visit through completion of the study. The Baseline for diary symptoms was the average of the last seven assessments prior to Randomization. Pooled SDs and LS means were calculated based on an ANOVA model.
Time Frame: Baseline through the Final Visit (Day 21)
Population: Efficacy analyses were based on all randomized participants (intent-to-treat principle) with at least some SABA follow-up information.
Measure: Least Squares Mean (Standard Deviation); unit: number of puffs of SABA
Arm/Group | Pleconaril | Placebo
Number analyzed (Participants) | 143 | 148
number of puffs of SABA
  Baseline (n=143, n=148) | 0.99 (2.43) | 0.81 (2.43)
  Change From BL to Day 1 (n=131, n=138) | 0.15 (2.37) | -0.15 (2.37)
  Change From BL to Day 2 (n=137, n=146) | 0.19 (3.75) | -0.16 (3.75)
  Change From BL to Day 3 (n=135, n=146) | 0.29 (3.17) | 0.03 (3.17)
  Change From BL to Day 4 (n=137, n=147) | 0.17 (2.01) | 0.23 (2.01)
  Change From BL to Day 5 (n=135, n=147) | 0.04 (1.86) | 0.27 (1.86)
  Change From BL to Day 6 (n=131, n=146) | -0.05 (1.45) | 0.12 (1.45)
  Change From BL to Day 7 (n=135, n=144) | 0.17 (1.88) | 0.19 (1.88)
  Change From BL to Day 8 (n=129, n=141) | -0.09 (1.63) | 0.06 (1.63)
  Change From BL to Day 9 (n=131, n=142) | -0.24 (1.76) | -0.14 (1.76)
  Change From BL to Day 10 (n=130, n=144) | -0.26 (1.76) | -0.14 (1.76)
  Change From BL to Day 11 (n=128, n=141) | -0.13 (1.92) | -0.05 (1.92)
  Change From BL to Day 12 (n=129, n=139) | 0.01 (2.38) | -0.12 (2.38)
  Change From BL to Day 13 (n=130, n=139) | 0.03 (3.05) | -0.14 (3.05)
  Change From BL to Day 14 (n=131, n=140) | 0.20 (3.08) | -0.07 (3.08)
  Change From BL to Day 15 (n=126, n=137) | 0.40 (4.12) | -0.11 (4.12)
  Change From BL to Day 16 (n=126, n=136) | 0.32 (2.45) | 0.26 (2.45)
  Change From BL to Day 17 (n=127, n=138) | -0.00 (2.13) | 0.01 (2.13)
  Change From BL to Day 18 (n=130, n=139) | -0.30 (2.07) | 0.07 (2.07)
  Change From BL to Day 19 (n=121, n=133) | 0.10 (2.25) | 0.11 (2.25)
  Change From BL to Day 20 (n=108, n=118) | 0.19 (2.15) | 0.39 (2.15)
  Change From BL to Day 21 (n=78, n=83) | 0.25 (1.76) | 0.11 (1.76)
  Change From BL to Final Day (n=143, n=148) | -0.05 (2.11) | 0.12 (2.11)
  Change From BL to Week 1 (n=142, n=148) | 0.15 (2.10) | 0.08 (2.10)
  Change From BL to Week 2 (n=139, n=146) | 0.06 (2.88) | -0.12 (2.88)
  Change From BL to Week 3 (n=135, n=145) | 0.08 (1.93) | 0.22 (1.93)
  Change From BL to Final Week (n=143, n=148) | 0.09 (1.90) | 0.21 (1.90)

10. Secondary Outcome: LS Mean Change From Baseline in Asthma-Related Sleep Interference
Description: Participants entered their asthma-related changes in sleep into an e-diary once daily (in the morning) beginning at the Screening Visit through completion of the study. Changes from Baseline in asthma-related sleep interference were determined using the following question: How did cold and asthma symptoms interfere with your sleep? The question was scored as follows: 0 = None, no interference with sleep at all, 1 = Mild, not annoying or troublesome, adequate amount of sleep, 2 = Moderate, interfered somewhat with sleep, woke up a few times, average sleep, 3 = Severe, substantially interfered with sleep, poor sleep. The Baseline for diary symptoms was the average of the last seven assessments prior to Randomization. Pooled SDs and LS means were calculated based on an ANOVA model.
Time Frame: Baseline through the Final Visit (Day 21)
Population: Efficacy analyses were based on all randomized participants (intent-to-treat principle) with at least some sleep follow-up information.
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pleconaril | Placebo
Number analyzed (Participants) | 146 | 153
units on a scale
  Baseline (n=146, n=153) | 0.12 (0.29) | 0.07 (0.29)
  Change From BL to Day 2 (n=141, n=152) | 0.06 (0.34) | 0.01 (0.34)
  Change From BL to Day 3 (n=140, n=152) | 0.02 (0.39) | 0.04 (0.39)
  Change From BL to Day 4 (n=141, n=151) | 0.00 (0.37) | 0.03 (0.37)
  Change From BL to Day 5 (n=138, n=152) | -0.01 (0.37) | 0.02 (0.37)
  Change From BL to Day 6 (n=135, n=151) | -0.02 (0.38) | 0.05 (0.38)
  Change From BL to Day 7 (n=136, n=149) | -0.05 (0.40) | 0.05 (0.40)
  Change From BL to Day 8 (n=137, n=147) | -0.06 (0.37) | 0.03 (0.37)
  Change From BL to Day 9 (n=136, n=148) | -0.04 (0.39) | -0.00 (0.39)
  Change From BL to Day 10 (n=136, n=149) | -0.02 (0.41) | -0.02 (0.41)
  Change From BL to Day 11 (n=135, n=148) | -0.03 (0.40) | -0.02 (0.40)
  Change From BL to Day 12 (n=135, n=146) | 0.01 (0.39) | -0.02 (0.39)
  Change From BL to Day 13 (n=134, n=146) | -0.04 (0.36) | -0.01 (0.36)
  Change From BL to Day 14 (n=133, n=146) | -0.04 (0.38) | -0.01 (0.38)
  Change From BL to Day 15 (n=132, n=142) | -0.01 (0.46) | 0.04 (0.46)
  Change From BL to Day 16 (n=129, n=138) | -0.03 (0.39) | 0.01 (0.39)
  Change From BL to Day 17 (n=127, n=141) | -0.01 (0.36) | -0.03 (0.36)
  Change From BL to Day 18 (n=131, n=145) | -0.03 (0.34) | -0.05 (0.34)
  Change From BL to Day 19 (n=129, n=144) | -0.03 (0.38) | -0.03 (0.38)
  Change From BL to Day 20 (n=123, n=133) | -0.06 (0.39) | 0.02 (0.39)
  Change From BL to Day 21 (n=107, n=121) | -0.04 (0.35) | 0.05 (0.35)
  Change From BL to Final Day (n=146, n=153) | -0.02 (0.43) | 0.04 (0.43)
  Change From BL to Week 1 (n=145, n=153) | 0.00 (0.27) | 0.03 (0.27)
  Change From BL to Week 2 (n=142, n=152) | -0.05 (0.33) | 0.00 (0.33)
  Change From BL to Week 3 (n=138, n=150) | -0.02 (0.35) | -0.01 (0.35)
  Change From BL to Final Week (n=146, n=153) | -0.03 (0.36) | -0.00 (0.36)

ADVERSE EVENTS:
Time Frame: AE data is reported from the time of randomization to the end of the Follow-up Period (Day 21). The Screening Period and Pre-Exposure Periods are not included in this time frame.
Arm/Group | Pleconaril | Placebo
Serious Adverse Events (participants affected / at risk) | 0/154 | 0/157
Other Adverse Events (participants affected / at risk) | 6/154 | 9/157
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pleconaril (N=154) | Placebo (N=157)
Headache (Nervous system disorders) | 6 (6) | 9 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees not to publish or publicly present any interim results

of the study without the prior written consent of the sponsor. The investigator further agrees to provide to the sponsor 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication that report any results of the study. The sponsor shall have the right to review and comment with respect to publications, abstracts, slides, and manuscripts.